CLINICAL TRIAL: NCT04422028
Title: Bioavailability of a Formulation of Desogestrel 0.075 mg Coated Tablets With Regards to the Marketed Reference Product
Brief Title: Bioavailability of Desogestrel 0.075 mg Tablets With Regards to Reference Product
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Laboratorios Andromaco S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: HP8824-01
Record Dates: First submitted 2020-06-04; First posted 2020-06-09 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-03

CONDITIONS: Bioequivalence
MeSH Terms: interventions — Desogestrel; Patents as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Desogestrel Test Product (Experimental): Participants received two tablets of the test formulation containing Desogestrel 0.075 mg. The tablets were taken with water and in a fasting condition.
  Interventions: Drug: Desogestrel 0.075 MG
- Desogestrel Reference Product (Active Comparator): Participants received two tablets of the marketed reference formulation containing Desogestrel 0.075 mg. The tablets were taken with water and in a fasting condition.
  Interventions: Drug: Desogestrel 0.075 MG

INTERVENTIONS:
Drug: Desogestrel 0.075 MG — Test Drug
  Other Names: Investigational Medicinal Product
  Arms: Desogestrel Test Product
Drug: Desogestrel 0.075 MG — Reference Product
  Other Names: Cerazette (Trademark)
  Arms: Desogestrel Reference Product

SUMMARY:
This Pivotal study investigated the bioavailability in women of 2 tablet formulations containing Desogestrel 0.075 mg. The Pivotal study was performed at a single site with 30 subjects. Participants took 2 tablets of the test product and reference product in 2 periods and 2 sequences (either test after reference or reference after test). There was a washout of 14 days between each study period.

DETAILED DESCRIPTION:
The primary objective of the study is to investigate the relative bioavailability of Desogestrel of 2 tablet formulations with Desogestrel 0.075 mg to demonstrate bioequivalence of both formulations in terms of rate and extent of absorption:

* Test Product: Product manufactured by Laboratorios Andrómaco S.A.
* Reference Product: Cerazette [Trademark], product of Merck Sharp and Dohme Ltda., Brasil.

The 90% confidence intervals for the intra-subject coefficient of variation (Test versus Reference Product) for the main pharmacokinetic parameters area under the plasma concentration-time curve from time zero to time t (AUC0-t) and from time zero to 72 hours (AUC0-72), and maximum plasma concentration (Cmax) for total metabolite etonogestrel was determined.

Participants were confined in the study site for approximately 36 hours during each study period (for 12 hours pre-dosing and for 24 hours post dosing) during which pharmacokinetic (PK) blood samples were obtained. 16 blood samples were taken up to 24 hours after the administration in each period. Participants returned to the site to provide additional blood samples at 48 h, and 72 h postdose.

The washout period between the two study periods was 14 days. The samples from each participant were analyzed with 2 methods of highperformance liquid chromatography-tandem mass spectrometry bioanalytical assays to quantify total Dienogest and Ethinyl estradiol in plasma.

The safety objective was to evaluate the tolerability of both formulations in women by collecting adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Non-pregnant and non-breastfeeding women
* Women of childbearing age with an acceptable form of contraception during the study
* 18 to 55 years old inclusive; BMI greater than or equal to 18.51 and less than or equal to 29.99
* Non-smoking or smoke only 3 cigarettes every 7 days
* With results of laboratory tests, electrocardiogram and chest radiography in normal and / or negative or abnormal ranges but without clinical relevance and declared suitable for study by the doctor after the physical examination
* Capable to understand the Informed Consent Form

Exclusion Criteria:

* Study site staff or sponsor staff or family members
* With history of drug and/or alcohol abuse
* Smokers more tan 3 cigarettes every 7 days
* Vitamin supplements intake 7 days prior to the administration of the medications under study
* Any recent change in eating habits or physical exercise
* Using of a pharmacological therapy (except over the counter medication use 7 days prior to the study)
* Hypersensitivity to the study drug or to other chemically related compounds, history of serious adverse reactions or hypersensitivity to any medication
* Use, during the 28 days prior to the start of the study, of medications known to alter liver enzyme activity
* Consumption of beverages or food containing grapefruit or pink grapefruit, within 7 days prior to each administration of the study medication and consumption of alcohol, caffeine or beverages or foods containing xanthines 24 hours before each administration of the study medication until the last sample of each period
* History of any significant cardiovascular disease
* Acute disease that generates significant physiological changes from the time of selection until the end of the study
* HIV, Hepatitis B and/or C positive
* Presence or history of thrombophlebitis, thrombosis or thromboembolic disorders, deep vein thrombosis, pulmonary embolism or known coagulopathy.
* Donation or loss of a significant volume (more than 100 mL) of blood or plasma or platelets during the 3 months prior to the start of the study
* Subjects who have participated in any type of clinical study during the 3 months prior to the start of the study
* History of any gastrointestinal surgery that could affect drug absorption
* Presence of fainting history or fear to blood collection

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2020-01-11 (Actual); Primary Completion 2020-01-11 (Actual); Study Completion 2020-01-28 (Actual)

PRIMARY OUTCOMES:
Total etonogestrel: area under the plasma concentration-time curve from 0 to 72 hours (AUC0-72). | From tablet intake and up to 72 hours after tablet intake.
  19 samples up to 72 hours will be taken after the administration in each period.
Total etonogestrel: area under the plasma concentration-time curve from 0 to time t (AUC0-t) | From tablet intake and up to 72 hours after tablet intake.
  19 samples up to 72 hours will be taken after the administration in each period.
Total etonogestrel: Maximum plasma concentration (Cmax) | From tablet intake and up to 72 hours after tablet intake
  19 samples up to 72 hours will be taken after the administration in each period.
Total etonogestrel: Time to achieve maximum plasma concentration (tmax) | From tablet intake and up to 72 hours after tablet intake
  19 samples up to 72 hours will be taken after the administration in each period.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director Study Director, Study Director — Laboratorios Andromaco
Locations (1):
- Innolab, Santiago, Chile

IPD SHARING:
Plan to Share IPD: No